CLINICAL TRIAL: NCT01264692
Title: A Multi-center, Double-blind, Randomized, Placebo- and Active-controlled, Parallel-group, Proof-of-concept Study to Evaluate the Efficacy, Safety, and Tolerability of 10 mg of ACT-280778 in Patients With Mild to Moderate Essential Hypertension
Brief Title: Essential Hypertension
Acronym: REDUCE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-067A201
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — isobutyric acid 2-(2-((3-(4,7-dimethoxy-1H-benzoimidazol-2-yl)propyl)methylamino)ethyl)-5-phenylbicyclo(2.2.2)oct-5-en-2-yl ester; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): ACT-280778
  Interventions: Drug: ACT-280778
- Treatment B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Treatment C (Other): Amlodipine
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: ACT-280778 — 10 mg once daily for 28 ± 2 days
  Arms: Treatment A
Drug: Placebo — Placebo oral capsules matching ACT-280778
  Arms: Treatment B
Drug: Amlodipine — 10 mg once daily for 28 ± 2 days
  Arms: Treatment C

SUMMARY:
The purpose of this study is to demonstrate the antihypertensive efficacy of once daily oral administration of ACT 280778 on DBP compared to placebo after 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 75 years (inclusive) at screening.
* Body mass index (BMI) between 18 and 35 kg/m2 (inclusive) and body weight at least 50 kg at screening and prior to enrollment.
* 12-lead ECG without clinically relevant abnormalities measured at screening.
* Clinical chemistry, hematology, coagulation, virus serology, and urinalysis test results not deviating to a clinically relevant extent from the normal range at screening.
* Signed informed consent in the local language prior to any study-mandated procedure

Exclusion Criteria:

* Mean SBP > 180 mmHg.
* Severe, malignant, or secondary hypertension.
* Episodes of hypertensive crisis or hypertensive emergency within 6 months prior to enrollment.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions considered to be of clinical significance.
* E6 Severe coronary artery disease indicated by myocardial infarction, percutaneous coronary intervention, or coronary artery bypass graft within the last 12 months prior to enrollment.
* Angina pectoris within 6 months prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in mean(c) trough(d) SiDBP | Baseline to day 28
  Change from baseline(b) to Day 28 (± 2 days) of Period 2 (Visit 7)in mean(c) trough(d) SiDBP.

SECONDARY OUTCOMES:
Change in mean trough SiSBP. | Baseline to Day 28
  Change from baseline to Day 28 (± 2 days) of Period 2 (Visit 7) in mean trough SiSBP.

CONTACTS AND LOCATIONS:
Overall Officials: Kasra Shakeri-Nejad, MD, PhD, Study Director — Actelion
Locations (18):
- Israel (11):
  - Clinical Investigative Site 4000, Afula
  - Clinical Investigative Site 1003, Ashkelon
  - Clinical Investigative Site 1008, Beersheba
  - Clinical Investigative Site 1004, Giv‘atayim
  - Clinical Investigative Site 1009, Holon
  - Clinical Investigative Site 1000, Jerusalem
  - Clinical Investigative Site 1006, Nazareth
  - Clinical Investigative Site 1007, Nazareth
  - Clinical Investigative Site 1005, Safed
  - Clinical Investigative Site 1010, Tel Aviv
  - Clinical Investigative Site 1012, Tel Litwinsky
- Serbia (7):
  - Clinical Investigative Site 3001, Belgrade
  - Clinical InvestigativeSite 3003, Belgrade
  - Clinical Investigative Site 4001, Belgrade
  - Clinical Investigative Site 3004, Belgrade
  - Clinical Investigative Site 3000, Niška Banja
  - Clinical Investigative Site 4002, Pančevo
  - Clinical Investigative Site 3002, Zemun